CLINICAL TRIAL: NCT03250637
Title: Meat and Fiber Intake and Interaction With Pattern Recognition Receptors (TLR1, TLR2, TLR4, and TLR10) in Relation to Colorectal Cancer in a Danish Prospective, Case-cohort Study
Brief Title: Diet, Genes and Colorectal Cancer - With Focus on Toll-like Receptor Polymorphisms
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Vibeke Andersen, Clinical Professor, University of Southern Denmark
Other Study IDs: 19-TLR
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Cancer
Keywords: Gene-environment interaction; Candidate gene; Western style diet; Toll-like receptors; Prospective study; Nested case-cohort
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from buffy coeats
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colorectal cancer cases: 1038 participants diagnosed with colorectal cancer from the Diet, Cancer and Health cohort.
  Interventions: Other: Observational
- Sub-cohort members: 1857 persons randomly selected within the full cohort at time of entry into the Diet, Cancer and Health cohort. These participants serve as controls for the colorectal cancer cases.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Information on diet, lifestyle, weight, height, medical treatment, environmental exposures, and other socio-economic factors were collected at enrolment using questionnaires and interviews

SUMMARY:
The aim of this study is to investigate the interaction between diet - primary meat and fiber - and polymorphisms in Toll-like receptors in relation to risk of colorectal cancer in a Danish prospective cohort.

DETAILED DESCRIPTION:
Meat and dietary fibers have been associated with increased and decreased risk of colorectal cancer (CRC), respectively. Toll-like receptors (TLRs) regulate intestinal immune response in a complex interplay between the mucosal epithelium and the microbiota and may therefore be important modulators of diet-induced CRC and interact with other inflammatory mediators.

The aim of the study is to investigate the association with functional TLR polymorphisms in relation to risk of CRC and their interaction with dietary factors. Additionally, interactions with previously studied polymorphisms in IL10, IL1B, PTGS2 and NFKB1 will be assessed in order to examine possible biological pathways in meat-induced CRC.

Data are retrieved from the Danish prospective "Diet, Cancer and Health" study encompassing 57,053 persons which were recruited between 1993 to 1997. Between 1994 and 31th December 2009, 1038 CRC cases has been diagnosed. A sub-cohort of 1857 persons has been randomly selected within the full cohort at time of entry into the cohort. The study design is a nested case-cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Born in Denmark and had no previous cancers at study entry

Exclusion Criteria:

* Previous or present cancer(s) at study entry

Ages: 50 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: The Diet, Cancer and Health study is an ongoing Danish cohort study designed to investigate the relation between diet, lifestyle and cancer risk. The cohort consists of 57,053 persons, recruited between December 1993 and May 1997. All the subjects were born in Denmark, and the individuals were 50 to 64 years of age and had no previous cancers at study entry. Blood samples, anthropometric measures and questionnaire data on diet and lifestyle were collected at study entry.
  The present study uses a nested case-cohort design. Follow-up is based on population-based cancer registries. Between 1994 and 31th December 2009, 1038 CRC cases were diagnosed. A sub-cohort of 1857 persons has randomly been selected within the full cohort at time of entry into the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 2895 (Actual)
Dates: Start 1993-12 (Actual); Primary Completion 1997-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Colorectal cancer | Between 1994 and 31th December 2009
  Follow-up was based on population-based cancer registries

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Andersen, MD, PhD, Study Director — University of Southern Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tjonneland A, Olsen A, Boll K, Stripp C, Christensen J, Engholm G, Overvad K. Study design, exposure variables, and socioeconomic determinants of participation in Diet, Cancer and Health: a population-based prospective cohort study of 57,053 men and women in Denmark. Scand J Public Health. 2007;35(4):432-41. doi: 10.1080/14034940601047986. PMID 17786808
- [Derived] Kopp TI, Vogel U, Tjonneland A, Andersen V. Meat and fiber intake and interaction with pattern recognition receptors (TLR1, TLR2, TLR4, and TLR10) in relation to colorectal cancer in a Danish prospective, case-cohort study. Am J Clin Nutr. 2018 Mar 1;107(3):465-479. doi: 10.1093/ajcn/nqx011. PMID 29566186
- See also: Description of the Diet, Cancer and Health cohort — http://www.cancer.dk/forskning/center-for-kraeftforskning/kost-gener-miljoe/kost-kraeft-helbred/